CLINICAL TRIAL: NCT06925490
Title: Clinical and Radiographic Evaluation of Pulpotomy Using 3Mixtatin Versus Pulpectomy Using Metapex in Vital Primary Molars Diagnosed With Symptomatic Irreversible Pulpitis in Children Aged 4 to 9 Years: A Randomized Clinical Trial.
Brief Title: Comparison of 3Mixtatin Pulpotomy and Metapex Pulpectomy in Primary Molars With Irreversible Pulpitis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nora Mohamed Mosaad Hussien, Pedodontist, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3Mixtatin and Metapex pulpitis
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Irreversible Pulpitis; Primary Teeth; Pulp Disease, Dental
Keywords: 3Mixtatin; irreversible pulpitis; metapex; pulpectomy; pulpotomy
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Metapex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metapex pulpectomy (Active Comparator): Single-visit pulpectomy using Metapex, . Calcium hydroxide-iodoform mixture (Metapex) is an ideal pulpal filling material for primary teeth.
  Interventions: Drug: Metapex
- 3Mixtatin Pulpotomy (Experimental): pulpotomy with 3 mixtatin (triple antibiotic paste of (Metronidazole, cefixime, and Ciprofloxacin mixed with simvastatin ) applied in the vital pulp therapy
  Interventions: Drug: 3Mixtatin

INTERVENTIONS:
Drug: Metapex — Pulpectomy using Metapex
  Arms: metapex pulpectomy
Drug: 3Mixtatin — pulpotomy treatment when applying 3mixture of antibiotic (Metronidazole, cefixime, and Ciprofloxacin) along with simvastatin
  Arms: 3Mixtatin Pulpotomy

SUMMARY:
The present study aims to evaluate the clinical and radiographic success of pulpotomy using 3Mixtatin versus pulpectomy using Metapex in primary molars with irreversible pulpitis in children aged 4 to 9 years.

DETAILED DESCRIPTION:
Primary teeth play an essential role in esthetics, phonatics, and mastication, that's why they should be preserved as the best space maintainers until their proper exfoliation time. Various pulp therapies were suggested based on the extent of carries, including vital pulp therapy (direct pulp capping, pulpotomy) and non-vital pulp therapy (pulpectomy). Current guidelines from the American Academy of Pediatric Dentistry (AAPD) and the British Society of Paediatric Dentistry (BSPD) recommend pulpectomy as the gold standard treatment for vital primary molars diagnosed with irreversible pulpitis. Pulpectomy is a non-vital treatment procedure where the entire pulp tissue is extirpated and the root canals debrided and shaped to receive a resorbable material to fill the canal space in the affected primary tooth.

In recent years, a paradigm shift has emerged towards performing pulpotomy, a more conservative approach that involves partial removal of the pulp tissue, furthermore, a previous histological study of teeth with irreversible pulpitis showed that inflammation and microbial invasion are confined to the coronal pulp, sparing the radicular pulp. This finding concurred that pulpotomy could represent a viable treatment option for teeth diagnosed with irreversible pulpitis, as it preserves tooth structure, enhances healing potential in the remaining pulp promoting long-term clinical and radiographic success.

Recently, the concept of a newer economical material "3Mixtatin" has come into research and has been studied for its use in direct pulp capping, inflammatory root resorption, and pulpotomy in primary teeth. The material is a combination of 3Mix (cefixime, metronidazole, and ciprofloxacin) and a statin (Simvastatin).

3Mixtatin, incorporates Simvastatin, an antihyperlipidemic drug, into the triple antibiotic paste, Simvastatin was used as an anti inflammatory and bioinductive agent, whereas 3Mix served as an antibacterial agent.

Statin components are emerging materials in regenerative dentistry. Evidence from both experimental and clinical studies supports the notion of 'pleiotropic' effects of statins, they improve osteoblasts function and suppress function of osteoclast leading to enhanced bone formation. Therefore, they might improve odontoblastic function resulting in improved dentin formation. Statins are also thought to induce angiogenesis and increase neuronal cell. Consequently, they play a role in pulp regeneration along with dentin regeneration. In addition, sufficient evidence exists in support of the potent anti-inflammatory properties of statins, they reduce circulating C-reactive protein (CRP) and pro-inflammatory cytokines, lowering the amount of interleukin-6 and interleukin-8 in inflamed pulpal tissues.

Owing to limited availability of data in researches and in order to reach conclusive results on whether pulpotomy can be offered as an alternate treatment to pulpectomy in vital primary molars diagnosed with irreversible pulpitis, our study aims to evaluate clinical and radiographic success of of pulpotomy using 3Mixtatin versus pulpectomy using Metapex with vital primary molars diagnosed with symptomatic irreversible pulpitis in children aged 4 to 9 years.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 4 to 9 years with vital primary molars showing signs of irreversible pulpitis.
* Children with spontaneous pain lasting a few seconds to several hours.
* Pain is intensified by thermal stimulus and persists after its removal.
* Pulp hemorrhage after performing access cavity and deroofing of pulp chamber showing reddish pink healthy pulp tissue.
* Radicular pulp health is verified by achieving hemostasis within eight minutes of compression using a cotton pellet with 5% sodium hypochlorite.
* Absence of peri-apical or inter-radicular radiolucency, widening of periodontal ligament space, internal or external root resorption.

Exclusion Criteria:

* Unrestorable primary molars.
* Primary molars with uncontrolled pulp hemorrhage or pulp necrosis.
* Medically compromised patients who have systemic disease.
* Uncooperative children who refuse treatment.
* Children whose parents are unwilling to place stainless steel crowns.
* Children whose parents or caregivers refuse to participate in the study or are unable to attend follow-up visits.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 3, 6, 9, and 12 months follow-up period
  * Pain to percussion will be assessed by applying a light-tapping force to the relevant tooth using the blunt end of the dental probe. Tapping will be applied as gently as possible from a 1 cm distance, either present or absent.
  * Swelling will be assessed through clinical examination, either present or absent.
  * The sinus tract or fistula will be assessed through clinical examination, either present or absent.
  * The mobility of teeth will be assessed by applying pressure to the ends of two metal instruments, either present or absent.
  * The principal investigator and the co-supervisor will undertake this clinical assessment on every recall visit during the 3, 6, 9, and 12 months follow-up period.

SECONDARY OUTCOMES:
Radiographic Success | 6 and 12 months
  * Radiolucency at the furcation or periapical area, internal or external root resorption, will be examined (present or not) through digital periapical radiographs.
  * The radiographic assessments will be performed as baseline data at the first visit following the procedure completion and at 6 and 12 months after the baseline
  * The Two blind assessors will independently evaluate the radiographic outcomes.
Post operative pain | 1 week, 3, 6, 9, and 12 months.
  After the completion of treatment, post-operative pain will be assessed using the Visual analog scale. This scale comprises six faces, with numbers ranging from 0 to 10 and word descriptions. During follow-up visits, the patients are asked to point to the face that best represents their feelings.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Ibrahim El Shahawy, Professor, Study Director — Professor of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University; Marwa Aly Fouad, Associate professor, Study Chair — Associate Professor of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University

IPD SHARING:
Plan to Share IPD: No